CLINICAL TRIAL: NCT02567123
Title: The Effects of Gait Retraining in Runners With Patellofemoral Pain: A Randomized Trial
Brief Title: Running Study for Runners With Chronic Knee Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not Applicable Clinical Trial.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNM-17714
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

ARMS (2):
- Experimental (Experimental): Runners are switched from a rearfoot strike running pattern to a forefoot strike running pattern.
  Interventions: Behavioral: Experimental
- Control (No Intervention): Runners continue to use their normal rearfoot strike running pattern with no intervention in place.

INTERVENTIONS:
Behavioral: Experimental
  Arms: Experimental

SUMMARY:
The purpose of this study is to determine whether changing foot strike pattern from a rearfoot strike to a forefoot strike reduces chronic running-related knee pain. It is believed that switching foot strike pattern from a rearfoot strike to a forefoot strike pattern will reduce associated running-related patellofemoral knee pain.

DETAILED DESCRIPTION:
Runners will come to the Gait Analysis Lab on north campus of the University of New Mexico, HSSB 168, for the first running trial. During this time you will fill out a health questionnaire, receive an assessment by a physical therapist, and be given a new pair of running shoes to use for the duration of the study.

Runners will be equipped with several reflective markers, which will be placed on your lower body. Runners will then complete several passes across a runway while we record your running with a motion analysis system. Runners will be equipped with a mouthpiece and nose clip. You will run for 10 minutes while we collect the gases you breathe.Twenty-four hours after you complete this running trial, you will come to our Exercise Physiology lab in Johnson Center, B143 to perform the training sessions. During this time you will run for about 10-30 minutes in front of a mirror and receive feedback from the research team. You will perform these training sessions eight times over two weeks. Twenty-four hours after your last training session, you will perform another follow-up running trial, which will be the same as the first trial. After completing the second running trial, you will be allowed to return to your normal running routine for about one month. After one month, you will return to the Gait Analysis lab to perform a final running trial, which will be the same as the first and second running trials.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of patellofemoral pain
2. No history of any cardiovascular issues.
3. Currently running as part of training program

Exclusion Criteria:

1. No patellofemoral pain present.
2. Not currently running as part of training program
3. Other lower extremity pain and/or injury that interferes with ability to run.
4. Pregnant
5. Not in the selected age ranges
6. Presence of cardiovascular or cardiopulmonary diseases

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pain | 6 weeks

SECONDARY OUTCOMES:
Knee abduction | 6 weeks
Knee range of motion | 6 weeks
ankle flexion | 6 weeks
ankle range of motion | 6 weeks
Knee flexion | 6 weeks
Patellofemoral Stress | 6 weeks
Patellofemoral contact force | 6 weeks
Achilles tendon force | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Mermier, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Relph N, Greaves H, Armstrong R, Prior TD, Spencer S, Griffiths IB, Dey P, Langley B. Running shoes for preventing lower limb running injuries in adults. Cochrane Database Syst Rev. 2022 Aug 22;8(8):CD013368. doi: 10.1002/14651858.CD013368.pub2. PMID 35993829
- [Derived] Roper JL, Harding EM, Doerfler D, Dexter JG, Kravitz L, Dufek JS, Mermier CM. The effects of gait retraining in runners with patellofemoral pain: A randomized trial. Clin Biomech (Bristol). 2016 Jun;35:14-22. doi: 10.1016/j.clinbiomech.2016.03.010. Epub 2016 Apr 7. PMID 27111879